CLINICAL TRIAL: NCT02780063
Title: The Effects of Dilation Medication on Lenstar Measurements for Cataract Surgery
Brief Title: Medications Effect on Lenstar Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15-00908
Record Dates: First submitted 2016-05-16; First posted 2016-05-23 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Cataract
Keywords: Dilation; Intraocular; Ophthalmology
MeSH Terms: conditions — Cataract; Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenstar Biometry (Experimental): Lenstar biometry will be performed on each eye prior to dilation. Subjects eyes will be dilated and subject will wait 20 minutes. Lenstar biometry will be performed after the 20 wait time.
  Interventions: Other: Lenstar Biometer

INTERVENTIONS:
Other: Lenstar Biometer — uses optical principles (laser interferometry) to measure axial length, measuring distance from the corneal apex to the retinal RPE. In addition to axial length, it also measures corneal thickness, anterior chamber depth, lens thickness, radii of curvature of flat and steep meridian, axis of flat meridian, white to white distance, and pupil diameter.

SUMMARY:
Prior to cataract surgery the lens must be calculated to appropriately fit a patient for the intraocular lens implant. Lenstar is an optical biometer that calculates the axial length, keratometry, lens thickness, pupillometry, and anterior chamber depth. Dilation drops are routinely used in eye exams in addition to pre-cataract surgery. The dilation drops include Tropicamide 1%, and Phenylephrine 2.5%. The Tropicamide achieves the dilation of the pupil which causes an anterior rotation of the ciliary body, which may affect the Lenstar measurements. This study is to determine if dilating medications affect the lens power prediction for emmetropia by the Lenstar biometer. Prior to dilation, Lenstar biometry will be performed on each eye. Patients will receive dilation medication and after waiting 20 minutes Lenstar biometry will be performed on each eye. Dilation and measurement with Lenstar will be done as standard of care. Measurements and calculations from before and after will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for cataract surgery undergoing routine evaluation of cataracts.

Exclusion Criteria:

* Patients that have had their cataracts removed
* Patients that cannot undergo routine evaluation for cataract surgery (because they are too ill to sit upright in a chair)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Baseline Lens Power will be compared to Post dilation measurements using Lenstar biometer | One Day

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ostrovsky, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States